CLINICAL TRIAL: NCT04433858
Title: An Open Label Study of the Safety and Efficacy of Psilocybin in Participants With Treatment-Resistant Depression (P-TRD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: COMPASS Pathways (Industry)
Responsible Party: Principal Investigator, Scott T. Aaronson, M.D, Director, Clinical Research Programs, Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14947563
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 25mg of Psilocybin
  Note: CA site only is re-dosing participants with an exacerbation in depressive symptoms at a minimum of 12 months post-initial dosing.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — open-label
  Other Names: COMP360

SUMMARY:
The primary objective of this study is to evaluate the efficacy of psilocybin (25 mg) administered under supportive conditions to adult participants with severe TRD, in improving depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least moderate Major Depressive Disorder (MDD)

Exclusion Criteria:

* Comorbidities

Note for CA site: Only Veterans are Eligible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | From Baseline (Day -1) to three weeks post-dose.
  MADRS is a clinician-rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity. Response = >50% decrease and Remission =< 10 actual score.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Aaronson, MD, Principal Investigator — Sheppard Pratt Health System
Locations (2):
- United States (2):
  - VA Palo Alto Healthcare System/Stanford Medicine, Palo Alto, California
  - Sheppard Pratt Health System, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellis S, Bostian C, Donnelly A, Feng W, Eisen K, Lean M, Conlan E, Ostacher M, Aaronson S, Suppes T. Long-term outcomes of single-dose psilocybin for U.S. military Veterans with severe treatment-resistant depression - 12-month data from an open-label pilot study. J Affect Disord. 2025 Nov 15;389:119655. doi: 10.1016/j.jad.2025.119655. Epub 2025 Jun 9. PMID 40499827
- [Derived] Ellis S, Bostian C, Feng W, Fischer E, Schwartz G, Eisen K, Lean M, Conlan E, Ostacher M, Aaronson S, Suppes T. Single-dose psilocybin for U.S. military Veterans with severe treatment-resistant depression - A first-in-kind open-label pilot study. J Affect Disord. 2025 Jan 15;369:381-389. doi: 10.1016/j.jad.2024.09.133. Epub 2024 Sep 27. PMID 39343309